CLINICAL TRIAL: NCT05550168
Title: Effect of Low-level Laser Therapy on Orthodontic Tooth Movement During Miniscrew-supported Maxillary Molar Distalization in Humans: A Single-blind, Randomized Controlled Clinical Trial
Brief Title: Effect of Low-level Laser Therapy on Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Beren Özsoy, DMD, Research assistant, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NearEastU-001
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Low Level Laser Therapy
Keywords: Accelerated orthodontic tooth movement; Biostimulation; Molar distalization; Humans
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: A clinical trial with experimental and control groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Laser group) (Experimental): The participants in the intervention group experienced a total of 7 session laser applications on their randomly determined molar region during the 12-week clinical trial period.
  Interventions: Device: Low Level Laser therapy
- Contralateral (Non-laser group) (No Intervention): Laser was not applied to the contralateral side of the intervention group (n=10) and the individuals in the control group (n=10); thus, no application was made to accelerate tooth movement
- Control (Non-laser group) (No Intervention): Laser was not applied to the contralateral side of the intervention group (n=10) and the individuals in the control group (n=10); thus, no application was made to accelerate tooth movement

INTERVENTIONS:
Device: Low Level Laser therapy — The participants in the intervention group experienced a total of 7 session laser applications on their randomly determined molar region during the 12-week clinical trial period.
  Arms: Intervention (Laser group)

SUMMARY:
The objective of this trial is to investigate the effect of low-level laser therapy (LLLT) on orthodontic tooth movement during maxillary molar distalization over 12-week observation period.

DETAILED DESCRIPTION:
The duration of orthodontic treatment may be prolonged depending on many factors such as the ratio of bone remodeling, the tooth anchorage, the type of applied mechanics, patient cooperation, and the necessity of keeping the applied forces during the treatment within physiological limits.1-7 Prolonged treatment might affect the psychosocial status of the patient and might lead to a decrease in the level of patient cooperation, and increase the risk of developing a pathological incident such as dental caries, periodontal diseases, alveolar bone resorption and root resorption due to insufficient oral hygiene.8-10 Increasing the intensity of the applied force in an attempt to accelerate tooth movement will cause closure of the blood vessels, and necrosis in the periodontal ligament, and will lead to inhibition of any cellular activity, which is also known as hyalinization.3-7 Various approaches such as local-systemic drug administration, mechanical-physical stimulations, and surgically-assisted approaches aimed at reducing the resistance of periodontal tissues against tooth movement and the effect of changing environmental factors have been developed to accelerate tooth movement and shorten the treatment period without increasing the intensity of the orthodontic force.2 LLLT (low-level laser therapy ) is one of the methods used for tooth movement therapy. Due to its non-invasive nature, safety, accessibility and bio-stimulating effects, LLLT is considered to be a promising tool for the future of dentistry.10 LLLT is currently being used to help speed up the ratio of bone formation in the suture after rapid maxillary expansion,18 reduce pain after orthodontic activation,19-21 and accelerate tooth movement19-32 in orthodontic clinical practices. In the literature, many of the experimental and clinical studies conducted to accelerate tooth movement by using the bio-stimulating effect of laser have demonstrated that tooth movement can be accelerated with LLLT.20-26 When compared with the previously mentioned approaches, no study has yet been found reporting any negative systemic effects of LLLT so far. It has been stated that there is a need for clinical trials to investigate the effects of non-invasive approaches that have the potential to accelerate tooth movement in different dentoalveolar regions.33 In this context, no previous study examined the effects of LLLT on maxillary molar distalization using a miniscrew-supported intraoral appliance. The aim of this study is to examine the contribution and effects of LLLT on orthodontic tooth movement during maxillary molar distalization using a miniscrew-supported intraoral appliance when compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal class I or mild class II malocclusion,

  * No untreated decayed teeth,
  * Normodivergent skeletal pattern,
  * Fully erupted maxillary first and second molars,
  * Male and female individuals between the ages of 16 and 22,
  * Extracted or congenitally missing maxillary third molars,
  * Non smoker,
  * No alveolar bone loss or periodontal disease,
  * Bilateral class II molar relationship,
  * Absence of crowding or spacing in the posterior region,
  * Adequate oral hygiene.
  * No drug usage that may have an impact on the biology of tooth movement (Example; Non-steroidal anti-inflammatory drugs- NSAIDS)

Exclusion Criteria:

* • Hypodivergent or hyperdivergent skeletal pattern,

  * Alveolar bone loss or periodontal disease,
  * Systemic illnesses that might affect bone metabolism,
  * Any drug use that may have an impact on the biology of tooth movement (Example; Non-steroidal anti-inflammatory drugs- NSAIDS),
  * Inadequate oral hygiene,
  * Unilateral class II molar relationship,
  * Smoker,
  * Severe class II skeletal malocclusion (ANB>7°),
  * Crowding or spacing in the posterior region,
  * Missing maxillary second molars,
  * Existence of maxillary third molars,
  * Having untreated decayed teeth.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Amount of maxillary molar distalization | 84 days after
  Measurements were made using miniscrew as a reference point. Digital measurements were made on Geomagic Studio 2014 software to evaluate the amount of maxillary molar distalization. All 3D digital model measurements were coded, and the same researcher carried out two separate measurements 1-week apart to increase the reliability of the measurements. Parallelism was ensured between the dental arch and the Y-axis on the side where the measurements would be made by guiding the models. The parallelism of the dental arch to the Y-axis was also assessed from the lateral view. The midpoint of the first miniscrew and the mesial edge of the maxillary first molar were marked in the occlusal view. Then the distance between the projections of these two reference points to the Y-axis was measured. The difference between the two consecutive measurements indicated the 3-week amount of distalization in T1, T2, T3 and T4. This procedure was applied on both sides of all 3D models

CONTACTS AND LOCATIONS:
Locations (1):
- Beren Özsoy, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozsoy B, Gulduren K, Kamiloglu B. Effect of low-level laser therapy on orthodontic tooth movement during miniscrew-supported maxillary molar distalization in humans: a single-blind, randomized controlled clinical trial. Lasers Med Sci. 2023 Feb 20;38(1):76. doi: 10.1007/s10103-023-03736-y. PMID 36807215